CLINICAL TRIAL: NCT04579588
Title: Understanding Immunity to the Flu Vaccine in COVID-19 Patients
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Sayantani B. Sindher, Associate Professor of Medicine, Stanford University
Other Study IDs: IRB-58356; 5U19AI057229-17 (NIH)
Record Dates: First submitted 2020-10-06; First posted 2020-10-08 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Corona Virus Infection; Flu Vaccine; Immunity
MeSH Terms: conditions — Coronavirus Infections; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample, stool sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- COVID-19 participants
  Interventions: Biological: Flu shot
- Control participants
  Interventions: Biological: Flu shot

INTERVENTIONS:
Biological: Flu shot — All participants will receive a single shot of the flu vaccine

SUMMARY:
The purpose of this study is to measure immunity to the flu vaccine over time in patients who have had COVID-19 and may have other medical conditions including obesity, type 2 diabetes, chronic fatigue, or long-term COVID-19 symptoms. Adults and children (age 9 to 64) who had been diagnosed with COVID-19 as well as controls without COVID-19 will be invited to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 9 through 64 years
* Diagnosed with COVID-19 at least 2 months prior enrollment
* Patients with or without obesity, diabetes, chronic fatigue and/or long term COVID-19 symptoms
* Patients without COVID-19 diagnosis for controls

Exclusion Criteria:

* Received the influenza vaccine less than 4 months ago
* Pregnant or lactating
* Patients with special risks attendant to venipuncture
* Use of immunomodulatory medications that may impact vaccine immune response per clinician's judgment
* Contraindication to the flu vaccine
* Immunodeficiency or autoimmune disease that may impact vaccine immune responses per clinician's judgement

Ages: 9 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adults (18-64 years) and children (9-17 years) diagnosed and not diagnosed (controls) with COVID-19 and who may have other medical conditions including long term COVID-19 symptoms, chronic fatigue, type 2 diabetes, and obesity.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2020-10-29 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Testing immunity to the flu vaccine over time | 1 week
Testing immunity to the flu vaccine over time | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Sayantani Sindher, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No